CLINICAL TRIAL: NCT00977990
Title: Amplification of Merkel Cell Polyomavirus From Skin Swab Specimens
Brief Title: Amplification of Merkel Cell Polyomavirus From Skin Swabs
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909219; 09-C-N219
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-19

CONDITIONS: Polyomavirus
Keywords: Skin Swab; Self-Sample

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

* Polyomavirus are DNA-based viruses that infect vertebrates, including humans. Most people are not harmed by polyomavirus infection, but people with compromised immune systems may be harmed by these viruses, and are at greater risk for developing certain types of rare cancers.
* A recently discovered virus called Merkel cell polyomavirus (MCV) is a type of skin infection commonly found in humans. By using skin swabs to collect MCV, researchers hope to develop a laboratory culture model of MCV for future research.

Objectives:

- To use skin swabs to collect samples of Merkel cell polyomavirus for future study.

Eligibility:

- Individuals 18 years of age and older who are employed in the National Cancer Institute's Laboratory of Cellular Oncology.

Design:

* Participants will wipe a cotton swab across their forehead and eyebrows, and break off the end of the swab into a microcentrifuge tube. This procedure will be performed after work hours.
* No other treatment or procedure will be given as part of this protocol.

DETAILED DESCRIPTION:
Polyomaviruses are a class of DNA-based viruses that infect vertebrates, including humans. A majority of humans are chronically infected with multiple polyomavirus types. In immunocompetent subjects, chronic polyomavirus infection is generally harmless. A recently-discovered virus called Merkel cell polyomavirus (MCV) is believed to chronically infect the skin of a substantial fraction of adult subjects. It has recently been shown that MCV DNA can be amplified from skin swab specimens using PCR methods. The goal of our study is to recover full-length (5.5 kb) MCV genomes from skin swab specimens taken from healthy laboratory volunteers. We will recombine any recovered MCV genomes and attempt to propagate them in cell culture. If successful, the work would provide the first laboratory culture model for MCV replication. The recombinant DNA work has received approval from the NIH Institutional Biosafety Committee

Our study population would be drawn from roughly two dozen co-workers in the Lab of Cellular Oncology's Building 37 Sections. LCO co-workers are an appealing study population because they are generally familiar with the biology of MCV. Candidate study participants will be reminded that, given the high prevalence of asymptomatic MCV infection among healthy adults, the detection of MCV DNA in skin swabs clearly cannot be construed as having any diagnostic, clinical or social significance.

Subjects who agree to participate in the study will wipe a cotton swab across their forehead and eyebrows. Study subjects will break off the end of the swab into a microcentrifuge tube. To avoid study participation during federal work hours, the specimen collection will be performed prior to or after the study subject's work shift. Each sample will be assigned a letter code. A key for the letter code will exist only in Dr. Buck's secure NCI server space.

Given the non-invasive nature of the sampling and the clear lack of potential harm arising from study participation, the proposal appears to be eligible for expedited review by the IRB's Special Studies section.

ELIGIBILITY:
* Study participants will be drawn from LCO co-workers in Building 37 Rooms 4106-4134. LCO members will be invited to participate without regard to gender, race, sexual orientation, or ethnic background.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-08-25; Study Completion 2010-05-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States